CLINICAL TRIAL: NCT03570489
Title: Randomized Controlled Study of the Effect of Cardiovascular Exercise in Uncontrolled Epilepsy: Efficacy, Side Effects and Quality of Life
Brief Title: Randomized Controlled Trial on Cardiovascular Exercise in Uncontrolled Epilepsy:
Acronym: Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit patients because of Covid 19 restrictions and because of lack of efficacy for primary endpoint
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFGBG-818131
Record Dates: First submitted 2018-05-28; First posted 2018-06-27 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2019-10

CONDITIONS: Refractory Epilepsy
Keywords: Cardiovascular fitness, refractory epilepsy,
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Open label randomized parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Use of an ergometric bicycle where patients will bicycle 5 Days a week for 20 minutes at a predetermine level
  Interventions: Behavioral: Exercise
- Relaxation (Sham Comparator): Patients will listen to a relaxation exercise involving muscle relaxation. This takes about 20 minutes and will be performed 5 Days/week
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Exercise — Patients will bicycle for 20 minutes per day for 5 days per week for 6 months
  Other Names: cardiovascular fitness
  Arms: Exercise
Behavioral: Relaxation — Patients will listen to a relaxation tape 20 minutes per day 5 Days a week for 6 months
  Arms: Relaxation

SUMMARY:
This is an open-label randomized controlled tria testing if an improvement in cardiovascular fitness can improve quality of Life and reduce seizure frequency in patients with refractory epilepsy.. Before the intervention each subject will undergo an evaluation of baseline cardiovascular fitness. Patients will be randomized into two groups One group will listen to a relaxation tape 5 days per week for 6 months and the other group will receive a ergometric cycle and perform a predetermined level of exercise per day , 5 days per week for 6 months. Randomization will be conducted an external randomization center based on a sequence of random numbers.

Changes in concomitant antiepileptic drugs (AED) treatment during the study will be minimized, and restricted to AED changes deemed to be necessary to address AED-related toxicity.

Medical examination; body weight; fitness test, including ECG and BP measurements, seizure frequency; adverse effects (unstructured interview); details of concomitant concomitant treatment, mood assessment by using the Hospital Anxiety and Depression Scale-Anxiety (HADS); health related quality of life (RAND-36), E4-data downloading, will be done at baseline and after 6 months

Primary endpoint: Proportion of patients with at least 50% seizure reduction

Secondary endpoints: Median percent reduction in seizure frequency, HADS score, RAND-36 score, fitness score; adverse events, changes in concomitant AED treatment, E4 data

.

DETAILED DESCRIPTION:
Objectives

The primary objective of this study is to assess the effect of a 6-month course of standardized physical exercise, added on to pre-existing stable AED treatment, on seizure frequency in patients with epilepsy aged 16 to 65.

Secondary objectives include the assessment of the effect of a 6-month course of standardized physical exercise, added on to pre-existing stable AED treatment, on (i) depressive and anxiety symptom scores; (2) health-related quality of life; (3) adverse

events.

Study design

Open-label randomized controlled trial. Before the intervention each subject will undergo an evaluation of cardiovascular fitness using the cycle ergometric test and his/her work level ((Wmax/kg) transformed into a stanine (1-9) score. Patients will be randomized into two groups by applying a stratification procedure which will allow a similar proportion of patients with high fitness (stanine score 5 to 9) and low fitness (stanine score 1 to 4) in both groups. Randomization will be conducted by telephone through an external randomization center based on a sequence of random numbers.

Of the two randomized groups, one (Intervention group) will receive a course of standardized physical exercise for at least 5 days per week while the other group (control group) will randomize to listening to a computerized disc (CD) on muscular relaxation..

Changes in concomitant AED treatment during the study will not be allowed unless for adverse events related to the AEDs.

Study procedures

Patients considered to be eligible for the study will undergo initially a 4-week prospective baseline to ascertain baseline seizure frequency. After confirming their eligibility based on seizure frequency recording, patients will be examined by a study physician and by a physical therapist who will conduct an ergonomic test with a stationary bicycle under ECG and blood pressure monitoring to determine the level of cardiovascular fitness required for stratification. Thereafter the patients will be randomized to the intervention and the control group.

The intervention group will receive a course of standardized physical exercise designed to fulfill the Swedish recommendations (FYSS) on exercise for disease-prevention (150 min per week of average intensity); at least 5 days per week for 6 months using a bicycle ergometer for 30 minutes a day. An individually adjusted workload will be determined by the physical therapist to achieve moderate intensity workout based on maximal oxygen uptake (VO2)max and percentage of maximal heart rate. Patients in the other group (control group) will be randomized to listen to a CD on muscular relaxation every day for 20 minutes and continue with their usual lifestyle. At enrollment, subjects randomized to the intervention group will be provided with a bicycle ergometer. requirements) as well parameters related to seizure activity.

The following evaluations will be conducted at the times indicated, which correspond to hospital visits:

Time 0 (enrollment): Medical examination; body weight; fitness test (Åstrand submax test, which is a submaximal test of aerobic fitness.), including ECG and BP measurements, seizure frequency (last 4 weeks); adverse effects (unstructured interview); details of concomitant concomitant treatment, mood assessment by using the Hospital Anxiety and Depression Scale-Anxiety (HADS); health related quality of life (RAND-36).

Month 1, 2, 3, 4 and 5: Seizure frequency (recorded daily on seizure calendars), adverse effects (unstructured interview); body weight; details of concomitant treatment, E4-data downloading, advice on exercise from physical therapist.

Month 6: Medical examination; body weight; fitness test, including ECG and BP measurements, seizure frequency; adverse effects (unstructured interview); details of concomitant concomitant treatment, mood assessment by using the Hospital Anxiety

and Depression Scale-Anxiety (HADS); health related quality of life (RAND-36), E4-data downloading,

Any additional testing (e.g. EEG, laboratory tests) may be performed as considered clinically indicated by the treating physician.

Sample size and statistical analysis

Assuming that 40% of patients in the intervention group vs. 20% of patients in the control group have a 50% or greater reduction in seizure frequency compared with baseline, 79 patients per group provide 80% power to identify a difference between groups at a significance level of 0.05. To account for potential dropouts, a total of 100 patients per group will be randomized.

The primary analysis will be intent-to-treat (ITT) using "The Last Observation Carried Forward " (LOCF) extrapolation when appropriate. Per-protocol analysis (PPT) will exclude patients discontinuing prematurely the study and patients with less than 75% compliance with exercise requirements.

Ethical aspects

The study protocol has been approved by the Ethics Committees of Gothenburg in behalf of the participating centers. Before the study, all patients will be informed about the objectives and implications of the study, and will be asked to sign an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years to 65 years
2. An established diagnosis of focal epilepsy
3. A frequency of at least 3 focal seizures (including focal to bilateral tonic-clonic) during a 4 week-prospective baseline, despite ongoing treatment with one to 4 AEDs
4. Stable AED treatment for at least 4 weeks, and no expected need to modify current AED treatment over the subsequent 6 months.
5. Capability to follow instructions (or has a caretaker who will help) and keep a seizure calendar
6. Ability to understand the purpose, procedures and potential risks and benefits associated with participation in the study;
7. Willingness to give freely written informed consent

Exclusion Criteria:

1. Any associated condition contraindicating non-competitive physical exercise
2. Patients already engaged in regular daily physical exercise program;
3. A history of seizures induced by exercise
4. A history of psychogenic non-epileptic seizures
5. Pregnancy or puerperium
6. Alcohol or substance abuse
7. Any condition (for example, an unstable or progressive medical condition) which, in the investigator's assessment, may interfere with the evaluation procedures or the objectives of the study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with at least 50% seizure reduction | Change from baseline at 6months
  Determined by seizure diary

SECONDARY OUTCOMES:
Change in anxiety and depression ratings | Change from Baseline at 6 months
  Reduction in Hospital Anxiety and Depression Scale (HAD) scores.The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3. A total score can be between 0 and 21 for either anxiety or depression. A lower score indicates less depression or anxiety: a cut-off point of 8/21 indicates the presence of anxiety or depression
Change in Health-Related Quality of Life | Change from Baseline at 6 months
  Improvement in "RAND-36 -Measure of Health Related Quality of Life" version called Item Health Survey (Version 1.0) score. There are 8 domains with 36 items in total. The eight health concepts are: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain and general health perceptions. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In a second step, items in the same scale are averaged together to create the 8 scale scores. Scores represent the percentage of total possible score achieved.
Reduction in adverse event reporting | Improvement from baseline at 6 months
  Subjective reporting by patient
Median percent change in seizure frequency | Change from Baseline at 6 months
  Seizure Counts by seizure diary

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Ben-Menachem, MD,PhD, Principal Investigator — University of Gothenburg, Department of Clincial Neuroscience, Sahlgrenska Academy
Locations (1):
- Elinor Ben-Menachem, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The plan is to share but we are uncertain just now as to how